CLINICAL TRIAL: NCT02424604
Title: Recurrency After Inguinal Herniorraphy With Bi-layer Mesh
Brief Title: Recurrency After Inguinal Herniorraphy With Bi-layer Mesh (BLM)
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jesper Magnusson, MD, Karolinska Institutet
Other Study IDs: EPN 2015/351-31/1
Record Dates: First submitted 2015-04-07; First posted 2015-04-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2016-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim The overall aim with this study is to improve outcome after inguinal hernia repair (IHR). It is not known today if a re-operation due to recurrence after bi-layer mesh IHR is more complicated than compared with the golden standard method.

Method This project is a registry study. The National hernia register (Svenskt bråckregister, SBR) which started in 1992 include data that cover nearly 100% of all the country's hernia operations.

Patient data are collected from SBR. Patients who at the time of surgery were between 18-75 years of age and operated on due to primary inguinal hernia with any of the two mentioned techniques between 1992-2012 are eligible

DETAILED DESCRIPTION:
Background Surgical repair for inguinal hernia is the most common surgical procedure in the world. Since the introduction of repair with mesh reinforcement, relapses have decreased significantly. Recurrence of inguinal hernia affects only 1-2% after inguinal hernia repair (IHR) [1] and is no longer considered to be a big problem. One problem is that a large proportion of patients undergoing surgery develop chronic pain from the surgical area [2-4]. New meshes, with new design and new materials are continuously being introduced, with the aim of reducing the incidence of chronic pain. One of the most common meshes in use today is the so-called "double-mesh" (bi-layer mesh) [1, 5]. Several studies have shown that bi-layer mesh can lead to some gains for the patient initially after surgery, but there is no scientific evidence available that suggest that bi-layer mesh is superior the traditional tension-free mesh repair in the long term [6, 7]. Several reports have shown that bi-layer mesh repair give results as good as the golden standard method, where a single sheet mesh is used.

The surgical technique differ somewhat with respect to which layer of the abdominal is being used [8], when using a bi-layer- or a single sheet mesh. With the bi-layer mesh you use the abdominal layer that is usually used (the pre-peritoneal space) in case of re-operation due to recurrence after open mesh repair. Re-operation after bi-layer mesh IHR is incompletely studied and it is unclear if this is a more difficult surgical procedure compared with re-operation for recurrence after standard IHR.

Aim The overall aim with this study is to improve outcome after IHR. It is not known today if a re-operation due to recurrence after bi-layer mesh IHR is more complicated than compared with the golden standard method.

Method This project is a registry study. The National hernia register (Svenskt bråckregister, SBR) which started in 1992 include data that cover nearly 100% of all the country's hernia operations.

Patient data are collected from SBR. Patients who at the time of surgery were between 18-75 years of age and operated on due to primary inguinal hernia with any of the two mentioned techniques between 1992-2012 are eligible.

Statistics Parametric and non-parametric statistical methods for descriptive analysis will be used for comparison within and between the groups. Students t-test.

Power calculation The primary outcome variable for this registry study is the prevalence of recurrence after bi-layer mesh IHR. This is incompletely mapped. There is no need of a power calculation because the material of the registry is very large and any relevant differences between the groups should easily be detected.

Gain of knowledge The results of the study could show that either method of IHR (eg bi-layer mesh) is less suitable in surgical repair of inguinal hernia, which could be troublesome for those patients who had surgery with the method.

ELIGIBILITY:
Inclusion Criteria:

* all patients in a national registry "inguinal hernia" who had had a relapse after inguinal surgery between 1992-2012

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patinets with relapse after inguinal hernia surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of recurrence | up to 30 days after surgery
  Recurrence rate for BLM in Inguinal hernia surgery

SECONDARY OUTCOMES:
Number of surgical methods (BML and Lichtenstein) | up to 30 days after surgery
  Surgical methods used in reoperation due to relapse after BML and Lichtenstein?

OTHER OUTCOMES:
Minutes, time of surgery | up to 30 days after surgery
  Surgery time due to relapse after BML and Lichtenstein
Number of complications | up to 30 days after surgery
  Complication due to relapse, after BML and Lichtenstein?

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Magnusson, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital, Stockholm, Sweden